CLINICAL TRIAL: NCT02155049
Title: Phase 3 Study of Treatment of Soft Tissue Expansion and Exophthalmos in Inactive Thyroid Eye Disease Patients Using Drops of Prostaglandin Analogues.
Brief Title: Treatment of Soft Tissue Expansion in Inactive Thyroid Eye Disease Patients Using Drops of Prostaglandin Analogues
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Maya Eiger, Medical Doctor, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED-01; Thyroid eye disease (Registry Identifier: Prostaglandin Analogues)
Record Dates: First submitted 2014-05-21; First posted 2014-06-04 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Thyroid Associated Ophthalmopathies
Keywords: TED; Prostaglandin Analogues
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prostaglandin Analogues (Experimental): The patients will receive a single daily drop of bimatoprost for six months.
  Interventions: Drug: bimatoprost 0.03%

INTERVENTIONS:
Drug: bimatoprost 0.03% — The patients will receive a single daily drop of bimatoprost for six months.
  Other Names: Lumigan (Allergan, Inc, Irvine, California)

SUMMARY:
Prostaglandin analogues eye drops are common and effective treatment for decreasing Intra-Ocular Pressure (IOP) in Glaucoma patients. A number of recently published case reports have documented periorbital fat atrophy following treatment by prostaglandin analogues. In this study the investigators want to use this side-effect of prostaglandin analogues for the treatment of orbital and periocular fat proliferation in inactive Thyroid eye disease (TED) patients, as a conservative substitute for surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Inactive TED (Clinical Activity Score below 3)
* Significant exophthalmos or orbital fat expansion.

Exclusion Criteria:

* Previous prostaglandin analogues treatment due to glaucoma
* Known prostaglandin analogues sensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Bimatoprost effect on soft tissue amount and exophthalmos in inactive TED patients. | 6 months
  To document the effect of bimatoprost treatment on the amount of soft tissue and exophthalmos in inactive TED patients. The following measurements will be performed pre, post and during treatment: orbital ultrasound (measuring the eyebrow fat, retro-orbicularis oculi fat and retrobulbar fat), Hertel exophthalmometry and Marginal Reflex Distance (MRD). The external appearance would be also documented by face picture.

SECONDARY OUTCOMES:
Number of participants with adverse events. | 9 months
  Determine the safety of bimatoprost treatment by estimating the probabilities of adverse outcomes. To estimate these probabilities we shall count the number of participants suffering from known side-effects of prostaglandin analogues such as increased eyelash growth and darkening of the periocular skin and iris; as well as any other side-effects observed during treatment.

OTHER OUTCOMES:
Bimatoprost effect reversibility after treatment cessation. | 3 months
  To measure the reversibility of bimatoprost treatment on the amount of soft tissue and exophthalmos at the end of the treatment course and 3 months post cessation. We shall perform the same measurements as described in the Primary Outcome section.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Eiger, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Ophthalmology clinics, Rabin Medical Center, Petah Tikva, Israel